

# TRIAL STATISTICAL ANALYSIS PLAN

c36049101-01

**BI Trial No.:** 1305-0016

**Title:** A phase I, open-label, non-randomized, single-dose, single-arm,

single-period study to investigate the metabolism and pharmacokinetics of [C-14]-labelled BI 1015550 after oral

administration in healthy male subjects

Final protocol (Version 1.0, c24519579-01)

Investigational

**Product:** 

BI 1015550

Responsible trial statistician:

Phone:

Fax:

Date of statistical

29-Jun-2021 SIGNED

analysis plan:

Version: 1

**** 

Proprietary confidential information

© 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | TABLE OF CONTENTS | |
|---|---|---|
| TITLE PA | AGE | 1 |
| 1. | TABLE OF CONTENTS | 2 |
| LIST OF | TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5.<br>5.1 | PRIMARY ENDPOINT | |
| 5.2 | SECONDARY ENDPOINTS. | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | 9 |
| 6. | GENERAL ANALYSIS DEFINITIONS | |
| 6.1<br>6.2 | TREATMENTSIMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | SUBJECT SETS ANALYSED. | |
| 6.5 | POOLING OF CENTRES | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | |
| 7.1<br>7.2 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINTS | |
| 7.4.1 | Primary analysis of the primary endpoints | |
| 7.5 | SECONDARY ENDPOINTS | |
| 7.5.1 | Key secondary endpoints | |
| <b>7.5.2</b> 7.5.2.1 | Secondary endpoints | |
| 1.3.4.1 | Secondary endpoint analysis | 1 / |
| 77 | EVTENT OF EVPOSUDE | 10 |

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| <b>7.8</b> | SAFETY ANALYSIS | 18 |
|--------------|-------------------------------------------|----|
| 7.8.1 | Adverse Events | 18 |
| <b>7.8.2</b> | Laboratory data | 19 |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | |
| 7.8.5.1 | Physical examination | 20 |
| 7.8.5.2 | Suicidality assessment (C-SSRS) | |
| 7.8.5.3 | Body weight | |
| 8. TIME | POINT OF RELEASE OF TREATMENT INFORMATION | 22 |
| 9. | REFERENCES | 23 |
| 11. | HISTORY TABLE | 25 |

# Boehringer Ingelheim TSAP for BI Trial No: 1305-0016 Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Analysis phases for statistical analysis of AEs, and actual treatment for | |
|---|---|---|
| | analysis of laboratory data and vital signs | 11 |
| Table 6.3: 1 | Subject sets analyzed. | 13 |
| | History table | |

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| $AUC_{0\text{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| BI | Boehringer Ingelheim |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| COVID | Coronavirus disease |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| ECG | Electrocardiogram |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPD | Important protocol deviations |
| LLOQ | Lower limit of quantification |
| MedDRA | Medical Dictionary For Regulatory Activities |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter analysis set |
| PR | Pulse rate |
| RAGe | Report appendix generator |
| RPM | Report Planning Meeting |
| SAE | Serious adverse event |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TS | Treated set |
| TSAP | Trial Statistical Analysis Plan |

# **Boehringer Ingelheim**

c36049101-01

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|------|-----------------------------|
| ULN | Upper limit of normal range |

# 3. INTRODUCTION

As per ICH E9 (1) the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary variables and other data.

This TSAP assumes familiarity with the CTP. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within Medidata Rave system.

| The statistical analyses will be performed within the validated working enviro | onment CARE, |
|---|---|
| including SAS <sup>TM</sup> (current Version 9.4, by | ), and a number |
| of SAS <sup>TM</sup> -based tools (e.g., macros for the analyses of AE data or laboratory Appendix Generator system (RAGe) for compilation/formatting of the CTR a | |
| PK parameters will be calculated using Phoenix WinNonlin <sup>TM</sup> software (version) | ion Phoenix 6.3 |

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in this TSAP are in accordance with the statistical methods described in the CTP.

# 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINT

Primary endpoint is as defined in Section 2.1.2 of the CTP:

# *Mass balance recovery of [C-14]-radioactivity*

• Amount of [C-14]-radioactivity excreted as a percentage of the administered single oral dose of BI 1015550 (C-14) in urine (fe<sub>urine, 0-12</sub>) and faeces (fe<sub>faeces, 0-12</sub>) as well as vomit (fe<sub>vomit, 0-12</sub>), if applicable.

#### 5.2 SECONDARY ENDPOINTS

# 5.2.1 Key secondary endpoints

Not applicable.

# **5.2.2** Secondary endpoints

Secondary endpoints are the following PK and safety endpoints as defined in Section 2.1.3 of the CTP.

PK endpoints of [C-14] BI 1015550, BI 1015550 and its metabolite BI 764333 in plasma:

- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

# Safety endpoint:

• Percentage of subjects with treatment emergent adverse events (TEAEs)





# 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on the treatment to be administered, and selection of dose, cf. Section 4 of the CTP.

Subjects will receive a single dose of [C-14]-labelled BI 1015550 as a 36 mL oral solution containing 18 mg BI 1015550 (17.16 mg unlabelled BI 1015550 mixed with 0.84 mg [C-14]-BI 1015550).

For statistical analysis of AEs, the following analysis phases are defined for each subject.

Table 6.1: 1 Analysis phases for statistical analysis of AEs, and actual treatment for analysis of laboratory data and vital signs

| Study analysis phase | Label | Start | End |
|---|---|---|---|
| Screening <sup>1</sup> | Screening | Date of informed consent | Date/time of administration of study drug |
| On treatment | BI 1015550 | Date/time of administration of study drug | Date/time of administration of<br>study drug + residual effect<br>period (7 days) |
| | | | or |
| | | | 12:00 a.m. on day after last contact date |
| | | | (whichever occurs first) |
| Follow-up | F/U | Date/time of administration of study drug + residual effect period (7 days) | 12:00 a.m. on day after last contact date |

<sup>&</sup>lt;sup>1</sup> See Section 6.7 for definition of baseline, which will be used in the statistical analyses of safety laboratory data and vital signs.

AE summary tables will present results for the on-treatment phase only. All AEs will be listed.

Safety laboratory data, vital signs and PK parameters will be analyzed with clear differentiation between baseline (cf. Section 6.7) and on-treatment measurements. Measurements will be considered on-treatment, if they were taken within the on-treatment phase as defined in Table 6.1: 1. Follow-up phase starts seven days after date/time of administration of the study drug since the residual effect period of the study drug is 7 days.

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an important PD (IPD). For definition of IPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (IPD)" (2) and the DV domain template.

If any IPDs are identified, they are to be summarised into categories and will be captured in the decision log. Categories which are considered to be IPDs in this trial are defined in the DV domain template. If the data show other IPDs, the definition in the DV domain template will be supplemented accordingly by the time of the Report Planning Meeting.

IPDs will be summarized and listed. Which kind of IPDs could potentially lead to exclusion from which analysis set is specified in the DV domain template. The decision on exclusion of subjects from analysis sets will be made at the latest at the Report Planning Meeting, after discussion of exceptional cases and implications for analyses.

Non-important COVID-19 related PDs will only be listed.

#### 6.3 SUBJECT SETS ANALYSED

The treated set (TS) and pharmacokinetic parameter analysis set (PKS) will be used as defined in the CTP, Section 7.3.

Table 6.3: 1 Subject sets analyzed

| | Subject set | |
|--------------------------------------|-------------|-----|
| Class of endpoint | TS | PKS |
| Disposition | X | |
| iPDs | X | |
| Primary endpoint | | X |
| Secondary PK endpoints | | X |
| Secondary safety endpoint | X | |
| Safety parameters | X | |
| Demographic/baseline characteristics | X | |
| Treatment exposure | X | |



#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one center.

# 6.6 HANDLING OF MISSING DATA AND OUTLIERS

**CTP**: "If a subject is removed from or withdraws from the trial prior to the administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after the administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF. In addition, the data will be included in the CRF and will be reported in the CTR."

**CTP**: "It is not planned to impute missing values for safety parameters."

One exception where imputation might be necessary for safety evaluation is AE dates. Missing or incomplete AE dates are imputed according to BI standards ( $\frac{3}{2}$ ).

Missing data and outliers of PK data are handled according to BI standards.

**CTP**: "Pharmacokinetic parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed."

# 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The last available value determined prior to study drug administration will be defined as baseline.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the Report Planning Meeting.

# 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (6).

The individual values of all subjects will be listed. Listings will be sorted by subject number, visit and planned time point (if visit/ planned time point is applicable in the respective listing). AE listings will be sorted by assigned treatment (see Section 7.8.1 below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters the following descriptive statistics will additionally be calculated:

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

# 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR. These will be based on the TS.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary. Concomitant non-drug therapies will be coded according to the most recent version of MedDRA.

Only descriptive statistics are planned for this section of the CTR.

**CTP:** Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

A medication will be considered concomitant, if it

- is ongoing at the time of study drug administration, or
- starts within the on-treatment phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM.

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analyzed as a specific endpoint. Any deviations from complete intake will be addressed in the Report Planning Meeting (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

# 7.4.1 Primary analysis of the primary endpoints

Only descriptive statistics are planned for this section of the CTR. These will be based on the PKS.

# Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

**CTP**: Plasma/urine concentration data and parameters of a subject which is flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses.

# Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic/ Pharmacodynamic Analyses of Clinical Studies" (4) and "Description of Analytical Transfer Files and PK/PD Data Files" (5).

#### 7.5 SECONDARY ENDPOINTS

# 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

# 7.5.2 Secondary endpoints

The analysis of secondary PK endpoints will be based on the PKS, the analysis of the secondary safety endpoint will be based on the TS.

# 7.5.2.1 Secondary endpoint analysis

**CTP:** The secondary endpoints will be calculated according to the BI SOP 001-MCS-36-476 (TMCP Data Analysis) and its reference documents and will be assessed statistically using the same methods as described for the primary endpoints.

Exclusion of PK parameters and exclusion of plasma concentrations are handled as described in Section 7.4.1.



#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report.

# 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trials" (7) and "Handling of missing and incomplete AE dates" (3).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to screening, on-treatment or follow-up phase as defined in <u>Section 6.1</u>. AEs will be analysed based on actual treatments, as defined in <u>Table 6.1: 1</u>.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of AESIs.

**CTP:** Hepatic injury is considered an AESI in this trial. A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase)  $\geq 3$  fold ULN combined with an elevation of total bilirubin  $\geq 2$  fold ULN measured in the same blood sample, or
- Aminotransferase (ALT, and/or AST) elevations  $\geq 10$  fold ULN

Furthermore, vasculitis is considered an AESI in this trial. Vasculitis is defined as any adverse event term included in the MedDRA SMQ Vasculitis (broad).

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (8), in addition to Deaths and Serious Adverse Events, 'other significant' AEs need to be listed in the clinical trial report. These will be any non-serious

adverse event that led to an action taken with study drug (e.g. discontinuation or dose reduced or interrupted).

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs and subjects with AESIs. AEs will also be summarized by maximum intensity.

The SOCs and preferred terms within SOCs will be sorted by descending frequency.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarized.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarized by treatment, primary SOC and preferred term.

# 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (9).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Unscheduled measurements of laboratory data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement. Descriptive statistics will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

Clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the Report Planning Meeting at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not.

Laboratory data will be compared to their reference ranges. Values outside the reference range as well as possibly clinically significant values will be highlighted in the listings. Possibly clinically significant laboratory values will be listed in Section 15.4.1.

Clinically relevant findings in laboratory data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analyzed as such.

# 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Unscheduled measurements of vital signs will be assigned to planned time points in the same way as described above for laboratory data. However, for vital signs, descriptive statistics will be calculated by planned time point based on the last value of the subject at that planned time point (or assigned to that planned time point). If the time of measurement is missing for a scheduled post-baseline measurement, the scheduled measurement will be used in calculation of descriptive statistics (as time difference between scheduled and unscheduled cannot be assessed).

If the time of measurement is missing for an unscheduled measurement, this measurement will be listed but will be ignored for the calculation of descriptive statistics.

Clinically relevant findings in vital signs data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analyzed as such.

# 7.8.4 ECG

Abnormal findings in ECG will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analyzed as such. No separate listing or analysis of ECG data will be prepared.

# **7.8.5** Others

### 7.8.5.1 Physical examination

Physical examination findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of physical examination findings will be prepared.

# 7.8.5.2 Suicidality assessment (C-SSRS)

Suicidality monitoring will be performed as described in Section 5.2.5.1 of the CTP. Results will only be listed, no further analysis will be prepared. Findings may also be reported as AEs as described in the CTP.

# 7.8.5.3 Body weight

Body weight will be analysed descriptively.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be loaded into the trial database at trial initiation.

#### 9. REFERENCES

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9; Note For Guidance on Design, Conduct, Analysis and Evaluation of Clinical Trials, current version |
|---|---|
| 2 | 001-MCS-40-413: "Identify and Manage Important Protocol Deviations (iPD)", current version; IDEA for CON |
| 3 | KM Asset BI-KMED-BDS-HTG-0035: "Handling of missing and incomplete AE dates", current version; KMED |
| 4 | KM Asset BI-KMED-TMCP-MAN-0014: "Noncompartmental PK/PD Analyses of Clinical Studies", current version; KMED |
| 5 | KM Asset BI-KMED-TMCP-MAN-0010: "Description of Analytical Transfer Files, PK/PD Data Files and ADA files", current version; KMED |
| 6 | KM Asset BI-KMED-BDS-HTG-0045: "Standards for Reporting of Clinical Trials and Project Summaries", current version; KMED |
| 7 | KM Asset BI-KMED-BDS-HTG-0066: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; KMED |
| 8 | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 9 | KM Asset BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", current version; KMED |

**Boehringer Ingelheim** 

c36049101-01

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1305-0016 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11. **HISTORY TABLE**

History table Table 11: 1

| Version | Date (DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 29-JUN-21 | | None | This is the final TSAP |